CLINICAL TRIAL: NCT07336849
Title: A Single-center, Prospective, Open Label Randomized Clinical Trial to Evaluate the Efficacy and Safety of Transcatheter Arterial Embolization Using 'Nexsphere-F' in Patients With Adhesive Capsulitis of the Shoulder Joint Refractory to Conservative Treatment.
Brief Title: Transcatheter Arterial Embolization Using Nexsphere-F for Chronic Shoulder Pain Refractory to Conservative Treatment
Acronym: TAE-FROST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Woosun Choi, Associate Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2505-006-641
Record Dates: First submitted 2025-12-15; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Adhesive Capsulitis of the Shoulder; Frozen Shoulder; Shoulder Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Transcatheter arterial micro-embolization (TAME) (Experimental): Participants assigned to the experimental group will undergo a one-time transcatheter arterial micro-embolization (TAME) procedure using Nexsphere-F. Usual conservative management for shoulder pain (e.g., physical therapy, analgesic medications, and/or intra-articular hyaluronic acid injection) may be provided as part of standard clinical care based on clinical judgement and patient preference and is not mandated by the study protocol.
  Interventions: Procedure: Transcatheter Arterial Micro- Embolization (TAME)
- Active Comparator: Usual care (conservative management) (Active Comparator): Participants assigned to the control group will not undergo transcatheter arterial micro-embolization (TAME) and will receive usual conservative management for shoulder pain as part of standard clinical care. Conservative treatments (e.g., physical therapy, analgesic medications, and/or intra-articular hyaluronic acid injection) may be provided based on clinical judgement and patient preference and are not mandated by the study protocol.
  Interventions: Other: Usual care (conservative management)

INTERVENTIONS:
Procedure: Transcatheter Arterial Micro- Embolization (TAME) — A one-time transcatheter arterial micro-embolization (TAME) procedure will be performed via radial artery access. After angiographic identification of abnormal neovascularity or hypervascular lesions associated with shoulder pain, target vessels will be superselected with a microcatheter and embolized using Nexsphere-F (gelatin-based bioresorbable embolic particles) until angiographic stasis or marked reduction of abnormal hyperemia is achieved, according to operator judgement.
  Arms: Experimental: Transcatheter arterial micro-embolization (TAME)
Other: Usual care (conservative management) — Usual conservative management for shoulder pain provided as part of standard clinical care. Conservative treatments (e.g., physical therapy, analgesic medications, and/or intra-articular hyaluronic acid injection) may be provided based on clinical judgement and patient preference and are not mandated or standardized by the study protocol.
  Arms: Active Comparator: Usual care (conservative management)

SUMMARY:
Evaluation of the efficacy and safety of transcatheter arterial embolization using 'Nexsphere-F' for pain relief in patients with adhesive capsulitis of the shoulder joint that does not respond to conservative treatment.

This study aims to investigate the efficacy and safety of transcatheter arterial embolization using embolic agents in patients with adhesive capsulitis of the shoulder joint. This is a single-center, prospective, open-label, randomized clinical trial.

DETAILED DESCRIPTION:
Evaluation of the efficacy and safety of transcatheter arterial embolization using 'Nexsphere-F' for pain relief in patients with adhesive capsulitis of the shoulder joint that does not respond to conservative treatment.

This study aims to investigate the efficacy and safety of transcatheter arterial embolization using embolic agents in patients with adhesive capsulitis of the shoulder joint. This is a single-center, prospective, open-label, randomized clinical trial.

Pain levels will be assessed via outpatient visits or telephone interviews at baseline (pre-procedure), and at 1 week, 1 month, 3 months, and 6 months post-procedure. During outpatient visits, the Visual Analog Scale (VAS), American Shoulder and Elbow Surgeons (ASES) score, Single Assessment Numeric Evaluation (SANE) score, shoulder range of motion (ROM), and the patient's subjective satisfaction (satisfied or not) will be recorded. Magnetic resonance imaging (MRI) of the shoulder joint will be performed both before the procedure and at 6 months post-procedure in both the control and intervention groups for comparative evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have voluntarily signed a written informed consent form after receiving an explanation of the purpose, methods, and potential effects of the clinical trial

  * Patients aged between 19 and 85 years

    * Patients with pain persisting for more than 3 months in the affected area and with a history of receiving physical therapy, analgesics/anti-inflammatory medications, or local injection treatments

      * Patients with a measured shoulder joint range of motion (ROM) of less than 90 degrees ⑤ Patients who agree not to receive any conservative treatment other than those permitted in this clinical trial (physical therapy, medication [NSAIDs, opioid analgesics, acetaminophen], intra-articular injections such as hyaluronic acid)

        * Patients who are willing to comply with the treatment and procedures of the clinical trial and participate in all follow-up evaluations through hospital visits or telephone surveys

Exclusion Criteria:

* Patients with a history of surgery on the shoulder joint targeted for the clinical trial prior to screening

  * Patients suspected of having a full-thickness rotator cuff tear

    * Patients with bleeding disorders or coagulopathies (e.g., idiopathic thrombocytopenic purpura, hemophilia, disseminated intravascular coagulation)

      * Patients with advanced atherosclerosis or vasospasm in the arm vessels, or those expected to have such conditions

        * Patients with a known hypersensitivity to gelatin

          ⑥ Patients with a known hypersensitivity to contrast media

          ⑦ Patients who are pregnant or breastfeeding

          ⑧ Patients with a localized infection at the pain site

          ⑨ Patients deemed inappropriate for participation by the investigator due to ethical concerns or potential impact on the clinical trial results

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) score | Baseline and 6 months after the procedure
  Change from baseline in shoulder pain severity assessed using the Visual Analog Scale (VAS) score, a 0-10 scale where 0 indicates no pain and 10 indicates the worst imaginable pain.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) scores at early follow-up | Baseline, 1 week, 1 month, and 3 months after the procedure
  Change from baseline in shoulder pain severity assessed using the Visual Analog Scale (VAS) scores, a 0-10 scale where 0 indicates no pain and 10 indicates the worst imaginable pain.
Shoulder joint range of motion (ROM) | Baseline, and at 1 week, 1 month, 3 months, and 6 months after the procedure
  Change from baseline in shoulder joint range of motion measured in degrees using a goniometer.
American Shoulder and Elbow Surgeons (ASES) score | Baseline and 6 months after the procedure
  Change from baseline in shoulder function assessed using the American Shoulder and Elbow Surgeons (ASES) Standardized Shoulder Assessment Form, a 0-100 scale where higher scores indicate better shoulder function.
Single Assessment Numeric Evaluation (SANE) | Baseline and 6 months after the procedure
  Change from baseline in shoulder function assessed using the Single Assessment Numeric Evaluation (SANE), a 0-100 scale where 0 represents complete disability and 100 represents normal shoulder function.
Patient satisfaction with treatment | 6 months after the procedure
  Patient satisfaction with treatment assessed using a 5-point Likert scale, where 1 indicates very dissatisfied and 5 indicates very satisfied.
Structural changes of the shoulder joint assessed by magnetic resonance imaging (MRI) | Baseline and 6 months after the procedure
  Structural changes of the shoulder joint assessed by magnetic resonance imaging (MRI), including the presence and severity of synovitis, capsular thickening, bone marrow edema, and tendon pathology, evaluated by qualitative and semi-quantitative radiologic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang Univerisity Hospital, Seoul, South Korea